CLINICAL TRIAL: NCT04144400
Title: Psychological Health in Military Personnel: Phase III
Brief Title: Psychological Health in Military Personnel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1432388-2
Record Dates: First submitted 2019-10-01; First posted 2019-10-30 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Well-being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRAVE Group (Experimental): The BRAVE program aims to examine the effectiveness of an intervention strategy designed to increase personal and work outcomes through the strengthening of quiet ego characteristics. The BRAVE intervention (delivered over four weeks) will ask study participants to use the app each week, with specific instructions on selecting one section each week and first listening to the longer version and reflect. At least two other times during the week they will be asked to listen to a recording of their choice on the same topic. On the final week (week 5) all participants (experimental and control) will return to the lab to complete post-study assessment tools (SART, post-study on-line questionnaire, provide a urine sample, and weight measurement).
  Interventions: Behavioral: Direction Check App
- Time Management Group (Active Comparator): The time management program aims to examine the effectiveness of an intervention strategy designed to increase personal and work outcomes through the strengthening of time management characteristics. The time management intervention (delivered over four weeks) will ask study participants to use the time management version of the app each week, with specific instructions on selecting one section each week and first listening to the longer version and reflect. At least two other times during the week they will be asked to listen to a recording of their choice on the same topic. On the final week (week 5) all participants (experimental and control) will return to the lab to complete post-study assessment tools (SART, post-study on-line questionnaire, provide a urine sample, and weight measurement).
  Interventions: Behavioral: Direction Check App (Time Management Version)

INTERVENTIONS:
Behavioral: Direction Check App — Direction Check is a simple, inexpensive app that builds resilience through balanced values to target the everyday personal and occupational stressors faced by military populations.
  Arms: BRAVE Group
Behavioral: Direction Check App (Time Management Version) — Direction Check (Time Management Version) is a simple, inexpensive app that builds resilience through time management exercises to target the everyday personal and occupational stressors faced by military populations.
  Arms: Time Management Group

SUMMARY:
The study is designed to compare the efficacy of a simple, non-spiritual, self-management strategy that can strengthen personal and occupational resources-resources that can positively impact adverse reactions to military-specific demands and promote personal and work outcomes. Our app-based intervention, designed to strengthen a balanced self-identity through affirmation of growth and balance values, will be adapted to military occupational contexts, utilizing an existing self-management strategy (QE) to a military occupational context to maximize it effectiveness in strengthening participants' balanced sense of self, which we expect to have positive benefit on personal and work outcomes in military service members.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study will include males and females between the ages of 17-70 years. Participants of all racial and ethnic backgrounds will be eligible to participate. Participants of all religious and spiritual orientations will be eligible to participate. Participants must be active-duty military personnel.

Exclusion Criteria:

* None.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-11 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Quiet Ego | Baseline, 5 weeks
  Change between baseline and five weeks, the Quiet Ego Scale (QES; Wayment, Bauer, & Sylaska, 2014) will be used to assess an identity that strikes a balance between a strong sense of agency (but not egoism) and a strong concern for the welfare of others. The QES is comprised of 14 items arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "I try to look at everybody's side of a disagreement before I make a decision" and "for me, life has been a continuous process of learning, changing, and growth." Higher scores on the QES indicate a stronger quiet ego. The QES has been found to have adequate internal validity (α = .76 to .78; (Wayment et al., 2014).
Self-Image | Baseline, 5 weeks
  The self-image and compassionate goals scale developed by Crocker and Canevello (2008) will be used to assess the change in self-image between baseline and five weeks. The scale is comprised of 13 items total with six items assessing self-image goals. The scale is arranged in a 5-point Likert-type format with responses ranging from 1 (Almost never) to 5 (Always). All items begin with the phrase, "In the past week, in the area of friendships, how much did you want to or try to..." Six of the items assess self-image goals such as, "get others to recognize or acknowledge your positive qualities" and "avoid taking risks or making mistakes." Higher scores for the self-image subscale represents a higher endorsement of self-image.
Compassioante Goals | Baseline, 5 weeks
  The self-image and compassionate goals scale developed by Crocker and Canevello (2008) will be used to assess the change in compassionate goals between baseline and five weeks. The scale is comprised of 13 items total with seven items assessing compassionate goals. The scale is arranged in a 5-point Likert-type format with responses ranging from 1 (Almost never) to 5 (Always). All items begin with the phrase, "In the past week, in the area of friendships, how much did you want to or try to..." Seven items asses compassionate goals such as, "be supportive of others" and "make a positive difference in someone else's life." Higher scores for the compassionate goals subscale represents a higher endorsement of compassionate goals.

SECONDARY OUTCOMES:
Spiritual Fitness | Baseline, 5 weeks
  Change between baseline and five weeks, the Spiritual Fitness Scale (SFS; Hammer, Cragun, & Hwang, 2013) will be used to assess the degree to which an individual has a sense of meaning, purpose, and accomplishment in their life that extends beyond the self (Peterson et al., 2011). The SFS is comprised of five items arranged in a 5-point Likert-type format with responses ranging from 1 (Not like me at all) to 5 (Very much like me). Sample items include: "I have a core of beliefs, ethics, and values that give my life a sense of meaning and purpose" and "The work I am doing in the military is meaningful to me." Higher scores on the SFS indicate a greater capacity to identify one's core self, access resources that facilitate the realizing of the core self and strivings, and experience a sense of connectedness with people and the world (i.e., spiritual fitness). The SFS has been found to have adequate internal consistency (α = .77; Hammer et al., 2013).
Positive and Negative Affect Schedule | Baseline, 5 weeks
  Change between baseline and five weeks, the positive and negative affect schedule (I-PANAS-SF; Thompson, 2007) will be used to assess positive and negative affect. The I-PANAS-SF is comprised of 10 items arranged in a 5-point Likert-type format with responses ranging from 1 (Very slightly or not at all) to 5 (Very much). Five items of the scale measure positive affect while the other five items measure negative affect. Respondents are asked to rate these positive and negative adjectives according to the extent to which each describes the way they have felt during the past week. Sample positive affect items include 'attentive', while sample negative affect items include 'upset'. Higher scores on both positive affect or negative affect indicate a tendency to experience a positive and negative mood. Both subscales (positive affect and negative affect) have been found to have adequate internal consistency (positive affect: α = .78; negative affect: α = .76; Thompson, 2007).
High Risk Demands | Baseline, 5 weeks
  Change between baseline and five weeks, a scale developed by Castro and Adler (2000) will be used to assess high-risk demands among respondents. The scale is comprised of seven items with short answer responses. Sample items include: "In the past week, how many hours of work have you average per day?" and "How many days have you been on a training exercise in the past 6 months?"
Traditional Occupational Demands | Baseline, 5 weeks
  Change between baseline and five weeks, the Organizational Constraints Scale (OCS; Spector & Jex, 1998) will be used to assess the ability of individuals to perform their jobs given their occupational demands. The OCS is comprised of 11 items arranged in a 5-point Likert-type format with responses ranging from 1 (Never) to 5 (Several times per day). Respondents are first asked to indicate how often it is difficult or impossible to do his or her job because of the listed items. Sample items include: "poor equipment or supplies," "inadequate training," and "interruptions by other people." Higher scores on the OCS indicate a high level of organizational constraints. The OCS has been found to have adequate internal consistency (α = .85; Spector & Jex, 1998).
Work Overload | Baseline, 5 weeks
  Change between baseline and five weeks, a shortened version of the overload subsection of the Michigan Organizational Assessment Questionnaire (MOAQ; Cammann, Fichman, Jenkins, & Klesh, 1983) will be used to assess work overload. The shortened MOAQ being utilized is comprised of three items arranged in a 7-point Likert-type format with responses ranging from 1 (Strongly disagree) to 7 (Strongly agree). Sample items include: "I never seem to have enough time to get everything" and "I have too much work to do to do everything well." One item is reverse-coded. Higher scores on the MOAQ and the overload subsection indicate greater work overload.
Coping | Baseline, 5 weeks
  Change between baseline and five weeks, the Emotion Regulation Questionnaire (ERQ; Gross, John, & Diener, 2003) will be used to assess participant's coping methods and ability among two common emotional regulation strategies - cognitive reappraisal and expressive suppression. The ERQ is comprised of 10 items total; six items which asses cognitive reappraisal and four items that assess expressive suppression. Each item is arranged in a 7-point Likert-type format with responses ranging from 1 (Strongly disagree) to 7 (Strongly agree). Sample items include: "When I want to feel more positive emotion (such as joy or amusement), I change what I am thinking about" and "I control my emotions by not expressing them." Higher scores in each subsection (reappraisal and suppression) indicate a higher tendency for respondents to use the related emotional regulation strategies. The ERQ has been found to have adequate internal consistency (α = .68 to .76; Gross et al., 2003).
Self-Compassion | Baseline, 5 weeks
  Change between baseline and five weeks, the Self-Compassion Scale (SCS; Raes, Pommier, Neff, & Van Gucht, 2011) will be used to assess the ability to extend compassion to the self. The SCS is comprised of 12 items and six subscales, each measuring a different component of self-compassion. Each item is arranged in a 5-point Likert-type format with responses ranging from 1 (Almost never) to 5 (Almost always). Sample items include: "When I fail at something important to me I become consumed by feelings of inadequacy" and "I try to see my failings as part of the human condition." Higher subscale scores on the SCS indicate greater endorsement of the related component of self-compassion. The SCS has been found to have adequate internal consistency (α = .86; Raes et al., 2011).
Family Functioning | Baseline, 5 weeks
  Change between baseline and five weeks, an adapted version of the Self-Report Measures of Family Functioning (SRMFF; Bloom, 1985) will be used to assess family functioning among two dimensions: family cohesion and family conflict. The SRMFF is comprised of 10 items total, five items relating to the dimension of cohesion and the other five items relating to the dimension of conflict. Respondents are asked to think about their family-life over the past week; each item is arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items relating to the dimension of cohesion include: "Family members really helped and supported one another" and "We really got along well with each other." Sample items relating to the dimension of conflict include: "We fought a lot in our family" and "Family members sometimes hit each other. Items 3 and 5 in both the dimensions of family cohesion and family conflict are reverse-coded.
Work-Family Conflict | Baseline, 5 weeks
  Change between baseline and five weeks, a shortened Work-Family Conflict Scale (WFSC; Carlson, Kacmar, & Williams, 2000) will be used to assess interrole conflict. The shortened WFSC being utilized is comprised of 12 items total; three items which assess time-based work interference with family, three items which assess time-based family interference with work, three items which assess strain-based work interference with family, and three items that assess strain-based family interference with work. Each item is arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). Sample items include: "My work keeps me from my family activities more than I would like" and "Due to stress at home, I am often preoccupied with family matters at work."
Personal Resources | Baseline, 5 weeks
  Change between baseline and five weeks, an adapted version of a social support and social strain survey developed by Wayment and Brookshire (2017) will be used to assess personal resources. The shortened version of the survey is comprised of six items arranged in a 5-point Likert-type format with responses ranging from 1 (Never) to 5 (All the time). Respondents are first asked to think about the "most important" person in their social network and are then asked about how often that person engaged in specific types of responses in the previous week. Sample items include: "listen to you when you wanted to talk". Higher scores for the social support questions indicate higher levels of social support. Higher scores for the social strain questions indicate higher levels of social strain. The survey has been found to have adequate internal consistency (social support: α = .89; social strain: α = .80; Wayment & Brookshire, 2017).
Military Pride | Baseline, 5 weeks
  Change between baseline and five weeks, three items adapted from a soldier will survey created by Marlowe, Furukawa, Griffith, Ingraham, and Kirkland (1985) will be used to assess military pride. The three items are arranged in a 5-point Likert-scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "I am proud to be in the Army" and "What I do in the Army is worthwhile." Higher scores on the survey indicate greater military pride.
Environment Life | Baseline, 5 weeks
  Change between baseline and five weeks, a scale developed by Huffman, Adler, Castro, and Dolan (2000) will be used to assess environmental life among respondents. The scale is comprised of five items arranged in a 5-point Likert-type format with responses ranging from 1 (Never) to 5 (Always). Sample items include: "I know what duty I will be doing day to day" and "I have a predictable mission schedule."

OTHER OUTCOMES:
Resilience to Adverse Events | Baseline, 5 weeks
  Change between baseline and five weeks, the Brief Resilience Scale (BRS; Smith et al., 2008) will be used to assess participant's resilience to adverse events. The BRS is comprised of six items total; three positively worded and three negatively worded. Each item is arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "I tend to bounce back quickly after hard times" and "I usually come through difficult times with little trouble." Items 2, 4, and 6 are reverse-coded. Higher scores on the BRS indicate greater resilience to adverse events. The BRS has been found to have adequate internal consistency (α = .93; Kyriazos et al., 2018).
Aggression | Baseline, 5 weeks
  Change between baseline and five weeks, a shortened version of the Aggression Questionnaire (AQ; Bryant & Smith, 2001) will be used to assess respondent aggression. The shortened AQ is comprised of 12 items arranged in a 5-point Likert-type format with responses ranging from 1 (Extremely uncharacteristic of me) to 5 (Extremely characteristic of me). Sample items include: "Given enough provocation, I may hit another person" and "My friends say that I'm somewhat aggressive." Higher scores on the AQ indicate greater levels of aggressive behavior. The AQ has been found to have adequate internal consistency (α = .53 to .80; Bryant & Smith, 2001).
Physiological-based stress | Baseline, 5 weeks
  Change between baseline and five weeks, to assess oxidative damage under resting (non-challenged) conditions, urinary excretion of oxidatively modified nucleic acids and lipids will be measured.
Sleep Disturbance | Baseline, 5 weeks
  Change between baseline and five weeks, two items adapted from the Pittsburgh Sleep Quality Index (PSQI; Buysee, Reynolds, Monk, Berman, & Kupfer, 1989) will be used to assess sleep disturbance. The first item asks participants: "On average how many hours of actual sleep do you get at night?". The second item asks, "During the past week, how would you rate your sleep quality overall?" and is arranged on a 4-point Likert-type format with responses ranging from 0 (Very good) to 3 (Very bad). The total PSQI has been found to have adequate internal consistency (α = .83; Smyth, 2012).
Perceived Stress | Baseline, 5 weeks
  Change between baseline and five weeks, a shortened Perceived Stress Scale (PSS; Cohen, Kamarck, & Mermelstein, 1983) will be used to assess the degree to which situations in one's life are appraised as stressful. The shortened PSS being utilized is comprised of 10 items arranged in a 5-point Likert-type format with responses ranging from 0 (Never) to 4 (Very often). Sample items include: "In the last week, how often have you felt that you were unable to control the important things in your life?" and "In the last week, how often have you been angered because of things that were outside your control?" Items 4, 5, 7, and 8 are reverse-coded. Higher scores on the PSS indicate greater appraisal of stressful life situations. The PSS has been found to have adequate internal consistency (α = .84 to .86; Cohen, Kamarck, & Mermelstein, 1983).
Symptoms/Reactions | Baseline, 5 weeks
  Change between baseline and five weeks, four items adapted from the Anger Rumination Scale (ARS; Sukhodolsky, Golub, & Cromwell, 2001) will be used to assess symptoms and reactions. The four items are arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "I thought about events that angered me for a long time" and "I thought about the reasons people treated me badly." Higher scores on the ARS indicate greater ruminative thoughts. The total ARS has been found to have adequate internal consistency (α = .93); Sukhodolsky et al., 2001).
Affective Commitment | Baseline, 5 weeks
  Change between baseline and five weeks, a shortened version of the Affective Commitment Scale (ACS; Meyer & Allen, 1984) will be used to assess commitment characterized by positive feelings of identification with, attachment to, and involvement in, the Army. The shortened version of the ACS that will be utilized is comprised of six items arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "I would be very happy to spend the rest of my career in the Army" and "The Army has a great deal of personal meaning for me." Items 3, 4, and 6 are reverse-coded. Higher scores on the ACS indicate a greater affective commitment to the army. The total ACS has been found to have adequate internal consistency (α = .87; Meyer & Allen, 1984).
Turnover Intentions | Baseline, 5 weeks
  Change between baseline and five weeks, in order to assess career intent, participants will be asked to respond to a single item which reads: "Which of the following best describes your career intentions at the present time?" Participants will respond to this question on a 5-point scale with responses ranging from 1 (Probably leave upon completion of my current obligation) to 5 (Definitely stay in until retirement, or longer).
Job Satisfaction | Baseline, 5 weeks
  Change between baseline and five weeks, four items adapted from a job satisfaction survey created by Quinn and Shepard (1974) will be used to assess the quality of military employment. The four items are arranged in a 5-point Likert-type format with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sample items include: "If a good friend of mine told me that he/she was interested in working in a job like mine I would strongly recommend it" and "Knowing what I know now, if I had to decide all over again whether to take my job, I would." Higher scores on the survey indicate greater job satisfaction.
Job Performance | Baseline, 5 weeks
  Change between baseline and five weeks, three items adapted from a job performance survey created by Griffin, Neal, and Parker (2007) will be used to assess individual task proficiency. The three items are arranged in a 5-point Likert-type format with responses ranging from 1 (Very little) to 5 (A great deal). Respondents are first asked to rate how often they have carried out a specific act over the past week. Sample items include: "Carried out the core parts of your job well" and "Ensured your tasks were completed properly." Higher scores on the survey indicate greater individual task proficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Huffman, PhD, Principal Investigator — Northern Arizona University

IPD SHARING:
Plan to Share IPD: No